CLINICAL TRIAL: NCT06500819
Title: Phase I Clinical Trial of Autologous B7-H3 Chimeric Antigen Receptor T Cells (B7-H3CART) in Children and Young Adults With Relapsed or Refractory Solid Tumor Expressing B7-H3 Target
Brief Title: Autologous B7-H3 Chimeric Antigen Receptor T Cells in Relapsed/Refractory Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Crystal Mackall, MD (Other)
Responsible Party: Sponsor-Investigator, Crystal Mackall, MD, Professor of Pediatrics and Medicine at Stanford University, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-74070; NCI-2025-00267 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Neuroblastoma; Sarcoma; Osteosarcoma
Keywords: Chimeric Antigen Receptor; Autologous T-Cells
MeSH Terms: conditions — Neuroblastoma; Sarcoma; Osteosarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lymphodepletion (Experimental): Fludarabine 30 mg/m2 per day IV for 4 days: 5, -4, 3, -2 Cyclophosphamide 500 mg/m2 per day IV for 3 days: -5, -4, -3 Subjects who meet cell infusion eligibility will receive IV B7-H3CART cells on Day 0.
  Interventions: Drug: B7-H3CART Dose (Intravenous)

INTERVENTIONS:
Drug: B7-H3CART Dose (Intravenous) — Subjects who meet cell infusion eligibility will receive IV B7-H3CART cells on Day 0.
  Dose level -1 (DL-1) 0.3 x 106 transduced T cells/kg
  Subjects who meet cell infusion eligibility will receive IV B7-H3CART cells on Day 0.
  Dose level 1 (DL1) 1 x 106 transduced T cells/kg
  Subjects who meet cell infusion eligibility will receive IV B7-H3CART cells on Day 0.
  Dose level 2 (DL2) 3 x 106 transduced T cells/kg
  Subjects who meet cell infusion eligibility will receive IV B7-H3CART cells on Day 0.
  Dose level 2 (DL2) 3 x 106 transduced T cells/kg
  Subjects who meet cell infusion eligibility will receive IV B7-H3CART cells on Day 0.
  Dose level 3 (DL3) 9 x 106 transduced T cells/kg

SUMMARY:
The purpose of this study is to test the manufacturing feasibility and safety of intravenous (IV) administration of B7-H3CART in children and young adult subjects with relapsed and/or refractory solid tumors expressing B7-H3 target using a standard 3+3 dose escalation design.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed malignant solid tumor (including neuroblastoma, soft tissue sarcoma, osteosarcoma, Ewing Sarcoma, and Wilms tumor) with evidence of incurable disease and tumor recurrence/progression after all available curative standard therapies.

   1. Subjects with neuroblastoma must have received or be intolerant to anti-GD2 antibody therapy.
   2. Subjects with Wilm's tumor must have received or be intolerant to ifosfamide or cyclophosphamide plus etoposide therapy or alternative salvage regimen.
   3. Subjects with embryonal rhabdomyosarcoma must have received or be intolerant to Adriamycin-based therapy.
   4. Subjects with surgically resected pulmonary osteosarcoma in first recurrence must have received surgical resection of metastatic nodules.
2. Subjects during dose escalation must have evaluable or measurable disease. Subjects during dose expansion must have measurable disease, except neuroblastoma which may have MIBG positive disease only.
3. B7-H3 positive expression on malignant cells is NOT required but archival tissue must be available, or the subject must be willing to undergo tissue biopsy for expression analysis.
4. Age: Must be ≥ 2 and ≤ 30 years of age.

   * For the first three subjects treated with B7-H3CART, must be ≥ 12 and ≤ 30 years of age.
5. Performance Status: Patients > 16 years of age must have Karnofsky ≥ 50%. Patients ≤ 16 years of age must have Lansky scale ≥ 50%; or ECOG performance status ≤ 2.
6. Prior Therapy

   1. No limit to the number of prior therapies.
   2. Prior Therapy Wash-out: At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy, which requires 5 half-lives. Radiation therapy must have been completed at least 3 weeks prior to enrollment, with the exception that there is no time restriction if the subject has measurable/evaluable disease outside the radiation port or the site of radiation has documented progression.
7. Normal Organ and Marrow Function (supportive care is allowed per institutional standards, i.e. filgrastim, transfusion)

   * ANC ≥ 750/uL*
   * Platelet count ≥ 75,000/uL*
   * Absolute lymphocyte count ≥ 150/uL*
   * Adequate renal, hepatic, pulmonary and cardiac function defined as:

     * Creatinine within institutional norms for age(i.e. ≤ 2 mg/dL in adults or according to table below in children <18 years) OR creatinine clearance (as estimated by Cockcroft Gault Equation) ≥ 60 mL/min

   Age (Years) Maximum & Serum Creatinine (mg/dL):

   Age (Years): ≤5 & Maximum Serum Creatinine (mg/dL): 0.8 Age (Years): 5 < age ≤ 10 Maximum Serum Creatinine (mg/dL): 1.0 Age (Years): >10-18 Maximum Serum Creatinine (mg/dL): 1.2 Age (Years): > 18 Maximum Serum Creatinine (mg/dL): 2.0
   * Serum ALT/AST ≤ 2.5x ULN (unless elevated ALT/AST is associated with disease involvement of the liver, in which case this criterion will be waived and not disqualify a patient).
   * Total bilirubin ≤ 1.5 mg/dl, except in subjects with Gilbert's syndrome.

     * Cardiac ejection fraction ≥ 45%, no evidence of physiologically significant pericardial effusion as determined by an ECHO,
     * No clinically significant ECG findings
     * No clinically significant pleural effusion
     * Baseline oxygen saturation > 92% on room air

       * if cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy); A subject will not be excluded because of pancytopenia ≥ Grade 3 if it is due to disease, based on the results of bone marrow studies.
8. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
9. Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four (4) months after receiving the preparative regimen or for as long as CART cells are detectable in peripheral blood.
10. Must provide informed consent. For subjects <18 years old, or adults with limited decision-making capacity, their legal authorized representative (LAR) (i.e. parent or guardian) must give informed consent. Pediatric subjects will be included in age appropriate discussion and assent will be obtained for those > 7 years of age, when appropriate. If a minor becomes of age during participation of this study, he/she will be asked to reconsent as an adult.

Exclusion Criteria:

1. Receiving any other current investigational agents.
2. History of other malignancy, except non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast), unless disease free for at least 3 years.
3. Presence of untreated brain metastases will be excluded. Subjects with previous CNS tumor involvement that has been treated and is stable for at least 3 months following completion of therapy are permitted. Patients who are clinically stable as evidenced by no requirements for corticosteroids, no evolving neurologic deficits, and no progression of residual brain abnormalities without specific therapy, are permitted.
4. Presence of fungal, bacterial, viral, or other infection that is uncontrolled. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
5. Ongoing infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti HCV positive) as the immunosuppression contained in this study will pose unacceptable risk. A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
6. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
7. Any medical condition that in the judgement of the sponsor investigator is likely to interfere with assessment of safety or efficacy of study treatment.
8. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
9. Pregnant females are excluded from this study because the effects of autologous B7-H3CART on the developing human fetus are unknown and because the chemotherapy agents used in this trial (cyclophosphamide and fludarabine) are category D agents with the potential for teratogenic or abortifacient effects. Additionally, because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with cyclophosphamide/fludarabine, breastfeeding should be discontinued if the mother is treated with cyclophosphamide/fludarabine. These potential risks may also apply to other agents used in this study.
10. Primary immunodeficiency or history of systemic autoimmune disease (e.g., Crohns, rheumatoid arthritis, systemic lupus) requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
11. Patients who require systemic corticosteroid or other immunosuppressive therapy. (A one-week washout from systemic corticosteroid or other immunosuppressive therapy is permitted.) Use of physiologic doses of corticosteroids (up to 3 mg/m2/day prednisone equivalent) are permitted. Use of topical, ocular, intra-articular, intra-nasal, or inhaled corticosteroids are permitted.
12. In the investigator's judgment, the subject is unlikely to complete all protocol required study visits or procedures, including follow up visits, or comply with the study requirements for participation.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of manufacturing autologous T cells | 2 years
  Feasibility of manufacturing autologous T cells transduced with Ef1a-CAR276 lentiviral vector expressing B7-H3 Chimeric Antigen Receptor (B7-H3-CART), using the Miltenyi CliniMACS Prodigy® system with dasatinib and protamine sulfate.
Safety and identify the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of a single dose of intravenous B7-H3CART | 2 years
  Assess the safety and identify the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of a single dose of intravenous B7-H3CART in children and young adults with relapsed and refractory solid tumors (i.e. soft tissue sarcoma, osteosarcoma, Ewing sarcoma, Wilms tumor, neuroblastoma) using the proposed dose escalation schedule.

SECONDARY OUTCOMES:
Clinical response in children and young adults | 2 years
  Assess clinical response in children and young adults with relapsed and refractory solid tumors treated with IV B7-H3CART.
Safety of B7-H3CART at the MTD/RP2D | 2 years
  Assess the safety of B7-H3CART at the MTD/RP2D in children and young adults with relapsed and refractory solid tumors treated with IV B7-H3CART.

CONTACTS AND LOCATIONS:
Overall Officials: Sneha Ramakrishna, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States